CLINICAL TRIAL: NCT04555993
Title: Comparison Between Ultrasound-Guided Transversus Abdominis Plane Block and Ultrasound-Guided Erector Spinae Plane Block in Postoperative Analgesia for Lower Abdominal Cancer Surgery. Randomised Double Blinded Control Study
Brief Title: Erector Spinae vs TAP in Lower Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Shaban Mohammed, Assistant lecturer of anesthesia and critical care medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-39-2019
Record Dates: First submitted 2020-09-01; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Pain
Keywords: erector spinae block; TAP Block; abdominal surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus abdomis plane block (Active Comparator): Patients will receive Transversus abdomis plane block
  Interventions: Procedure: lower abdominal surgery; Other: Transversus abdominis plane block
- Erector spinae plane block (Experimental): Patients will receive Erector spinae plane block.
  Interventions: Procedure: lower abdominal surgery; Other: Erector spinae plane block

INTERVENTIONS:
Procedure: lower abdominal surgery — Patients will undergo lower abdominal surgery under general anesthesia.
Other: Erector spinae plane block — patients will receive erector spinae plane block using 20 mL levobupivacaine (0.25%).
  Arms: Erector spinae plane block
Other: Transversus abdominis plane block — patients will receive transversus abdominis plane block using 20 mL levobupivacaine (0.25%).
  Arms: Transversus abdomis plane block

SUMMARY:
The aim of this study is to compare the analgesic effect and safety profile of erector spinae plane block with transverses abdominis plane block in controlling peri-operative pain for lower abdominal cancer surgery.

DETAILED DESCRIPTION:
Pain triggers a complex biochemical and physiological stress response leading to impairment of pulmonary, immunological and metabolic functions. Opioids are the current gold standard drug for postoperative pain relief, however exposure to large doses lead to multiple side effects of varying significance such as nausea, vomiting, dizziness, constipation, respiratory depression, hypoventilation and sleep breathing disorders. Therefore strategies other than opioids are recommended without sacrificing proper and effective analgesia. Especially in cancer patients who are more susceptible to tolerance and addiction.

The Transversus Abdominis Plane (TAP) block, is a regional anaesthesia technique used effectively in laparotomies. Unilateral analgesia to the skin, muscles, and parietal peritoneum of the anterior abdominal wall will be achieved without affecting visceral pain, when the anterior rami of the lower six thoracic nerves (T7-T12) and the first lumbar nerve (L1) are blocked.

Erector spinae plane block (ESPB) was shown to be an effective analgesic option for different types of surgeries. It's relatively a simple block, drug is injected in the plane between the erector spinae muscle and the vertebral transverse process. Blocking the ventral and dorsal rami of spinal nerves on the paravertebral area distributed from T2-T4 to L1-L2 and gives good coverage to visceral pain. Owing to the lower risk of blood vessel damage and neural damage compared to the epidural or the paravertebral block.

Both blocks haven't been compared to each other in this type of surgery before.

ELIGIBILITY:
Inclusion Criteria:

* Physical status ASA II.
* Age ≥ 18 and ≤ 65 Years.
* Cancer patients undergoing laparotomies for radical cystectomy or radical hysterectomy or low anterior resection (lower abdominal procedures).
* Patient is able to provide a written informed consent.
* Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.

Exclusion Criteria:

* Age <18 years or >65 years.
* BMI <20 kg/m2 and >40 kg/m2.
* Known sensitivity to local anaesthetics and morphine.
* History of psychological disorders and/or chronic pain.
* Significant liver or renal insufficiency.
* Contraindication to regional anaesthesia e.g. local sepsis, preexisting peripheral neuropathies and coagulopathy.
* Patient refusal.
* Severe respiratory or cardiac disorders.
* Pregnancy.
* ASA III-IV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours
  The total amount of morphine which was consumed post-operatively measured in milligrams

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption. | intraoperative
  The total amount of fentanyl which was consumed during the surgery measured in milligrams

OTHER OUTCOMES:
Postoperative nausea and vomiting | 24 hours postoperative
  the number of patients who had nausea and vomiting
Time for first rescue analgesia. | 24 hours postoperative
  the time at which the patient will request an analgesic
Heart rate | 24 hours
  the number of heart beats in one minute
Numerical rating scale for pain assessment. | 24 hours
  This is a numerical rating scale for pain assessment which ranges from 0 to 10 with the least pain at scale 0 and the worst pain at scale 10
mean arterial blood pressure | 24 hours
  the mean arteiral blood pressure measurend in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: waleed hamimy, Professor, Study Chair — Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

REFERENCES:
- [Background] Randerath WJ, George S. Opioid-induced sleep apnea: is it a real problem? J Clin Sleep Med. 2012 Oct 15;8(5):577-8. doi: 10.5664/jcsm.2162. No abstract available. PMID 23066371
- [Background] Finnerty O, Carney J, McDonnell JG. Trunk blocks for abdominal surgery. Anaesthesia. 2010 Apr;65 Suppl 1:76-83. doi: 10.1111/j.1365-2044.2009.06203.x. PMID 20377549
- [Background] Hebbard P. Subcostal transversus abdominis plane block under ultrasound guidance. Anesth Analg. 2008 Feb;106(2):674-5; author reply 675. doi: 10.1213/ane.0b013e318161a88f. No abstract available. PMID 18227342
- [Background] Yarwood J, Berrill A (2010). Nerve blocks of the anterior abdominal wall, Continuing Education in Anaesthesia Critical Care & Pain, Vol10, Issue 6, pp 182-186.
- [Background] Abrahams MS, Horn JL, Noles LM, Aziz MF. Evidence-based medicine: ultrasound guidance for truncal blocks. Reg Anesth Pain Med. 2010 Mar-Apr;35(2 Suppl):S36-42. doi: 10.1097/AAP.0b013e3181d32841. PMID 20216023
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539
- [Background] De Cassai A, Marchet A, Ori C. The combination of erector spinae plane block and pectoralis blocks could avoid general anesthesia for radical mastectomy in high risk patients. Minerva Anestesiol. 2018 Dec;84(12):1420-1421. doi: 10.23736/S0375-9393.18.13031-8. Epub 2018 Jul 9. No abstract available. PMID 29991225